CLINICAL TRIAL: NCT02776566
Title: Patient-Centered Anticoagulation Self-Monitoring in Minority Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, Edith A. Nutescu, Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2015-1193; K23HL112908 (NIH)
Record Dates: First submitted 2016-03-28; First posted 2016-05-18 (Estimated); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Thromboembolism; Blood Coagulation Disorders; Cardiovascular Disease; Vascular Disease
Keywords: Anticoagulation; Anticoagulation Management; Self-Testing; Self-Management; Warfarin; Thromboembolism; Blood Coagulation Disorders; Health Disparities; Minorities; African American; Hispanic; Cardiovascular Disease; Models of Anticoagulation Care; Tele-Health; Home Self-Testing
MeSH Terms: conditions — Thromboembolism; Blood Coagulation Disorders; Cardiovascular Diseases; Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anticoagulation Clinic (Active Comparator): Usual care through pharmacist managed anticoagulation clinic
  Anticoagulation Clinic (control): subjects will have their INR tested in clinic monthly (or more frequently if clinically indicated) via the Coaguchek® point-of-care device (which is the standard of care in the Anticoagulation Clinic) and receive dosing instructions and standardized education related to warfarin by a clinical pharmacist who provides care in the Anticoagulation Clinic.
  Interventions: Other: Patient Self-Monitoring vs Anticoagulation Clinic
- Patient Self-Monitoring (Experimental): In home self-monitoring and pharmacist guided education
  Patient Self-Monitoring (intervention): entails 3 education sessions of 90-120 minutes each (week 0, week 2, week 4): 2 provided on site in clinic and 1 in the patient's home, during which, self-testing competency and barriers and facilitators to self-monitoring will be evaluated. Subjects will follow with weekly (or sooner, if clinically indicated) in-home self-monitoring and follow-up weekly phone calls over 6 months by clinical pharmacists to guide warfarin dosing and reinforce key educational messages.
  Interventions: Other: Patient Self-Monitoring vs Anticoagulation Clinic

INTERVENTIONS:
Other: Patient Self-Monitoring vs Anticoagulation Clinic — Patient Self-Monitoring (intervention): entails 3 education sessions of 90-120 minutes each (week 0, week 2, week 4): 2 provided on site in clinic and 1 in the patient's home, during which, self-testing competency and barriers and facilitators to self-monitoring will be evaluated. Subjects will follow with weekly (or sooner, if clinically indicated) in-home self-monitoring and follow-up weekly phone calls over 6 months by clinical pharmacists to guide warfarin dosing and reinforce key educational messages.
  Anticoagulation Clinic (control): subjects will have their INR tested in clinic monthly (or more frequently if clinically indicated) via the Coaguchek® point-of-care device (which is the standard of care in the Anticoagulation Clinic) and receive dosing instructions and standardized education related to warfarin by a clinical pharmacist who provides care in the Anticoagulation Clinic.

SUMMARY:
The purpose of this study is to demonstrate the feasibility and effectiveness of anticoagulation self-monitoring coupled with an educational intervention in a minority underserved population.

DETAILED DESCRIPTION:
Despite favorable results and enhanced patient convenience, the adoption of patient self-monitoring for anticoagulation therapy has been limited primarily to non-minority and higher socioeconomic status individuals. While effectiveness has been studied, the factors influencing the adoption of self-monitoring of anticoagulation in minorities with the most barriers to accessing quality care in specialized clinics, are not known.

Hypothesis: Patient centered education and training intervention for minority patients will result in effective adoption of self-monitoring of anticoagulation therapy, resulting in anticoagulation control of comparable quality to that seen in specialized anticoagulation clinic-based monitoring.

The research objective of this proposal will be accomplished through 3 specific aims:

1. Identify patient and provider factors that influence adoption of anticoagulation self-monitoring in a minority population.
2. Adapt and refine an education intervention that both addresses identified barriers and emphasizes identified positive influences to anticoagulation self-monitoring.
3. Demonstrate the feasibility and effectiveness of anticoagulation self-monitoring coupled with an educational intervention in a minority population.

ELIGIBILITY:
Inclusion Criteria:

* > 21 years of age
* African American or Hispanic
* English speaking
* Has been on warfarin therapy > 3 months
* Plan to be on warfarin therapy > 12 months
* Willing ( or caregiver be willing) to do self-monitoring
* Willing to be randomized

Exclusion Criteria:

* Lack of access to a telephone
* Moderate to severe dementia (if lacks caregiver)
* Severe hearing impairment ( if lacks caregiver)
* Blindness ( if lacks caregiver)
* Life expectancy < 6 months
* Antiphospholipid antibody syndrome

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2016-01; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Percent time in therapeutic range (TTR) | Month 1, Month 2, Month 4, Month 7
  TTR will be calculated for each patient using the linear interpolation method. This method has been associated with clinical outcomes such as risk for thromboembolic events, and thus was selected over other methods of expressing the TTR such as fraction of International Normalized Ratio (INR) in range and cross-section of files

SECONDARY OUTCOMES:
Treatment Related Quality of Life | Baseline, Month 1, Month 7
  It will be evaluated using a 25 item validated questionnaire that assesses limitations, hassles, and positive impact with a Cronbach alpha for each of 0.87, 0.88 and 0.78 respectively
Anticoagulation Related Knowledge | Baseline, Month 1, Month 7
  It will be measured with an instrument containing 29 items at different levels of difficulty to allow differences in patient knowledge to be evaluated and has a person reliability coefficient of 0.75.
Adherence with Monitoring | Month 1, Month 2, Month 4, Month 7
  It is defined as the INR test completed within 24 hours of scheduled time and measured via the Coaguchek® device in home or clinic.
Self-Testing Competency (Intervention group only) | Baseline to 7 months
  It is defined as the ability to attain an INR reading and provider observed technique.
Self-Testing Accuracy (Intervention group only) | Baseline to 7 months
  It is defined as the concordance of self-reported and device-stored INR measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Edith A Nutescu, PharmD, MS, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided